CLINICAL TRIAL: NCT06579599
Title: Study on the Preventive Effect of Establishing an Integrated Working Group of Doctors and Nurses in Operating Room on Incision Infection in Orthopedic Surgery and Its Clinical Enlightenment
Brief Title: Study on the Preventive Effect of Establishing an Integrated Working Group of Doctors and Nurses in Operating Room
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: KY-2024-143
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Orthopedic Disorder; Incision Infection
Keywords: Orthopedic Disorder; Incision Infection; Operating room; Integration of medical staff
MeSH Terms: conditions — Musculoskeletal Diseases; Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine operating room nursing (No Intervention): Routine nursing interventions were put into practice in the operating room for the control group.
- an integrated working group nursing (Experimental): Received intervention through the establishment of an integrated working group comprising medical staff in the operating room.
  Interventions: Other: an integrated working group nursing

INTERVENTIONS:
Other: an integrated working group nursing — (1) Establishment of an integrated team in the operating room; (2) Development of a nursing plan; (3) Nursing safety training and reflection in the operating room; (4) Designate a person to manage instruments and equipment in the operating room and establish protocols (5) Nurses should also participate in the development of the patient's individualized surgical plan communicate with the surgeon about the preparation of items needed for surgery to ensure seamless coordination. Assist anesthesiologists and surgeons and oversee the implementation of aseptic procedures.
  Arms: an integrated working group nursing

SUMMARY:
To explore the preventive effect and clinical enlightenment of establishing an integrated working group of doctors and nurses in operating room on incision infection in orthopedic surgery.

DETAILED DESCRIPTION:
Surgery is the most used treatment in orthopedics. During orthopedic surgery, the integrity of the skin barrier is compromised, resulting in direct exposure of sterile tissue to the external environment and the potential impact of surgical instruments on local tissue. Additionally, orthopedic surgery procedures often entail prolonged duration, extensive surgical areas, and significant blood loss, all of which contribute to an elevated risk of surgical site infections. However, there are some limitations in the practical application of the conventional nursing model in the operating room. Against this backdrop, numerous new nursing models have emerged to meet contemporary demands. Among them, the integration of medical and nursing staff (MANS) in the operating room has garnered significant attention. Presently, this integrated model is predominantly employed in critical care settings and for postoperative infection prevention. However, the establishment and effectiveness of an integrated working group comprising both MANS in the operating room remains in its nascent stage of exploration, warranting further investigation into its clinical impact and implications.

ELIGIBILITY:
Inclusion Criteria:

* (1) All selected cases met the relevant diagnostic criteria outlined in the orthopedic disease guidelines. Diagnosis was confirmed through imaging methods.

  (2) The patients ranged in age from 18 to 70. (3) All individuals underwent surgery in the orthopedic department of our hospital.

  (4) The vital signs of the patients were essentially stable. (5) Patients possessed normal cognitive function before the operation and demonstrated the ability to listen, speak, read, and write.

Exclusion Criteria:

* (1) Orthopedic patients with multiple injuries in other locations (such as craniocerebral trauma, chest trauma, etc.); (2) Patients with severe internal diseases, such as severe anemia, severe diabetes, liver insufficiency; (3) Patients with chronic infectious diseases; (4) Patients with malignant tumor; (5) Patients with pathological fracture, such as bone tumor; (6) Patients with mental diseases and cognitive impairment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Incision infection rate | One month after surgery
  Incision infection rate = the number of postoperative incision infection / the total number of cases × 100%

SECONDARY OUTCOMES:
Incision recovery | On the 1 day of discharge
  On the day of discharge, the effect of incision healing was evaluated by the doctor and recorded by the nurse, including excellent: the surgical incision basically healed without adverse reactions; good: poor healing, mild redness, swelling and induration around the incision, but no suppuration; poor: the incision has been infected and suppurate. Excellent and good rate = (excellent + good) cases / total cases × 100%
Nursing quality | On the 1 day of discharge
  The nursing quality management questionnaire of operating room made by our hospital was used, and the quality control department staff or head nurse made an unannounced visit to evaluate the nursing quality
Adverse nursing risk events | On the 1 day of discharge
  the total adverse nursing risk rate of the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Feng Huang, BA, Principal Investigator — The Fourth Affiliated Hospital of Zhejiang University School of Medicine
Locations (1):
- The Fourth Affiliated Hospital of Zhejiang University School of Medicine, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No